CLINICAL TRIAL: NCT06315803
Title: Randomized Controlled Clinical Study to Validate the Clinical Accuracy and Safety of Biplanar Ultrasound-guided Puncture of Lumbar Interforamen in Adults
Brief Title: Randomized Controlled Clinical Study of Biplanar Ultrasound-guided Puncture of Lumbar Interforamen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Mao (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Yi Mao, clinician, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ChinaPLAGH20230601
Record Dates: First submitted 2024-03-05; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Lumbar Disc Herniation; Percutaneous Endoscopic Lumbar Discectomy; Three-dimension Ultrasound; Learning Curves
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Masking Description: There are practical differences in operation and blind methods cannot be achieved.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xplane ultrasound group (Experimental): The lumbar interforamen puncture was performed under the guidance of Xplane ultrasound with a X6-1 volume transducer probe (frequency range 1-6MHz, center frequency 3.2MHz).
  Interventions: Device: Real-time 3D Xplane ultrasound
- radiography group (No Intervention): The lumbar interforamen puncture was performed under the guidance of radiography with Mobile X-ray Image System (Arcadis Orbic 3D, Siemens, Germany) .

INTERVENTIONS:
Device: Real-time 3D Xplane ultrasound — After the puncture needle is in the skin, the longitudinal section of the Xplane mode can be adjusted to keep the needle in the proposed plane.
  Arms: Xplane ultrasound group

SUMMARY:
The goal of this clinical trial is to compare Xplane ultrasound with radiography for guidance of lumbar interforamen puncture in patients with lumbar disc herniation. The main question[s] it aims to answer are:

* The feasibility that the Xplane ultrasound assists surgeon in mastering lumbar interforamen puncture faster than radiography.
* The clinical accuracy and safety of the Xplane ultrasound-guidance lumbar interforamen puncture faster.

Participants will undergo lumbar interforamen puncture with guidance of Xplane ultrasound or radiography. If there is a comparison group: Researchers will compare the first success rate, number of punctures, number of radiographies, puncture time and operator confidence score.

ELIGIBILITY:
Inclusion Criteria:

1. 16 to 80 years of age;
2. symptoms and confirmatory signs of lumbar radiculopathy that persisted for at least 6 weeks;
3. LDH at a corresponding level and side on imaging;
4. surgical candidates for epidural steroid injection (ESI) or percutaneous endoscopic lumbar discectomy (PELD). If the patient underwent ESI and PELD surgery on the same day, we only selected the data for the first one.

Exclusion Criteria:

1. other diseases affecting the spine (tumor, infection, metabolic disease, immune system disease and fractures);
2. body mass index (BMI) greater than 32 kg/m2;
3. pregnancy;
4. refusal to participate;
5. severe mental illnesses in the trial.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
the first success rate | during operation
  the incidence of success on the first puncture of the target
number of punctures | during operation
  number of punctures of the target
number of radiographies | during operation
  number of radiographies during punctures
puncture time | during operation
  how long hands are in contact with the needle

SECONDARY OUTCOMES:
operator confidence score | Immediately after puncture
  operator confidence score
operative time | Immediately after surgery
  The time between the start of the surgery and the end of the surgery
incidence of puncture relevant complications | The patient was examined for neurovascular injury immediately after the puncture. Other complications were observed 1 month after surgery
  neurovascular injury, cauda equina syndrome, dural tear, injection, hematoma and organ injury
satisfaction of patients | 1 month after surgery
  satisfaction of patients(1-5points) from the last follow-up

OTHER OUTCOMES:
visual analog scale of pain | The day before surgery and 1 month after surgery
  pain scores (1-10) on the visual analog scale for waist and leg
Oswestry disability index | The day before surgery and 1 month after surgery
  Oswestry disability index
modified Macnab criteria type | the last follow-up (at least 1 month after surgery)
  modified Macnab criteria type (excellent,good,fair,poor)

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li YY, Liu YH, Yan L, Xiao J, Li XY, Ma J, Jia LG, Chen R, Zhang C, Yang Z, Zhang MB, Luo YK. Single-plane versus real-time biplane approaches for ultrasound-guided central venous catheterization in critical care patients: a randomized controlled trial. Crit Care. 2023 Sep 23;27(1):366. doi: 10.1186/s13054-023-04635-y. PMID 37742018
- [Result] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Result] Zhang M, Yan L, Li S, Li Y, Huang P. Ultrasound-guided transforaminal percutaneous endoscopic lumbar discectomy: a new guidance method that reduces radiation doses. Eur Spine J. 2019 Nov;28(11):2543-2550. doi: 10.1007/s00586-019-05980-9. Epub 2019 May 13. PMID 31087164